CLINICAL TRIAL: NCT02305693
Title: Comparison Between Letrozole and Laparoscopic Ovarian Drilling in Women With Clomiphene Resistant Polycystic Ovarian Syndrome (PCOS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sub 7
Record Dates: First submitted 2014-11-26; First posted 2014-12-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Active Comparator): 70 women will receive Letrozole (Femara®, Novartis, Switzerland) 2.5mg twice daily for 5 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding
  Interventions: Drug: Letrozole
- Ovarian drilling (Active Comparator): 70 women will have LOD in which the ovaries will be stabilised by grasping the ovarian ligament and monopolar diathermy will be used to do 4-10 punctures in each ovary. The number of punctures will be individualised according to the size of the ovary.
  Interventions: Procedure: Laparoscopic ovarian drilling

INTERVENTIONS:
Drug: Letrozole
  Arms: Letrozole
Procedure: Laparoscopic ovarian drilling
  Arms: Ovarian drilling

SUMMARY:
140 women with clomiphene resistant PCOS will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Letrozole, group 2 will have laparoscopic ovarian drilling (LOD).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in reproductive age, with an incidence of 5 -10%. Classically clomiphene citrate (CC) is the first approach to induce ovulation in patients with PCOS. Although 70-80% of PCOS women can ovulate by the treatment with CC, only 40%of the PCOS women become pregnant. Women who do not ovulate with increasing doses of CC are described as being CC-resistant and remain a major challenge in gynecologic endocrinology. Traditional alternatives for CC-resistant patients include gonadotropin therapy and laparoscopic ovarian diathermy.

Letrozole is an orally-active aromatase inhibitor, with good potential for ovulation induction. Letrozole acts by reducing estrogen production by blocking androgens to estrogens conversion. Additionally, it has no adverse effect on endometrium and cervical mucus (4). This releases the pituitary from negative feedback of estrogens and releases FSH. Also, an added positive effect is increased follicular sensitivity to FSH through amplification of FSH receptor gene expression.

Laparoscopic ovarian drilling (LOD) can avoid or reduce the need for gonadotropins for ovulation induction. Several potential mechanisms of action of LOD have also been suggested. The reduction of inhibin production following LOD is followed by an increase in FSH secretion and recruitment of a new cohort of follicles. Other theory is restoration of normal production of the putative gonadotropin surge after laparoscopic ovarian electrocautery. Moreover, drainage of androgens and inhibin from follicles surface may inhibit the excessive collagenisation of overlying ovarian cortex and facilitate Softening of ovarian tunica. Neighbouring follicles that are not undergoing atresia may then mature and gain access to the ovarian surface, facilitating ovulation. Initiation of normal inhibin B pulsatility by LOD appears to correlate with the postoperative onset of ovulatory cycles.

The main drawbacks of LOD are adhesions formation and ovarian atrophy. That is why minimising the number of diathermy points and avoiding diathermy near the ovarian hilum are recommended.

All women with clomiphene resistant PCOS attending the subfertility clinic of Cairo university hospitals will be invited to participate in the study. PCOS diagnosis will be based on chronic anovulation and sonographic picture of polycystic ovaries. Clomiphene resistance will be defined as failure of ovulation in spite of receiving 150mg of clomiphene citrate for 5 days starting from the 3rd-5th day of the menstrual cycle.

Exclusion criteria are age >40 years, other causes of infertility, hyperprolactinaemia, previous Letrozole or LOD therapy, and body mass index (BMI)>35.

The study will be explained to all the participants and a written informed consent will be obtained before participation.

Full history will be taken followed by complete examination and sonographic evaluation. Sonographic picture of polycystic ovaries will be defined when there are at least 12 follicles 2-9mm in the ovary and/or ovarian volume>10cm3 140 women with clomiphene resistant PCOS will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive Letrozole, group 2 will have LOD and group 3 will act as the control group with no intervention.

Group 1 will receive Letrozole (Femara®, Novartis, Switzerland) 2.5mg twice daily for 5 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. Group 2 will have LOD in which the ovaries will be stabilised by grasping the ovarian ligament and monopolar diathermy will be used to do 4-10 punctures in each ovary. The number of punctures will be individualised according to the size of the ovary.

Serial vaginal ultrasound scans were done starting from the 10th day of menstruation, the frequency of monitoring will be individualized according to the women's response. When the dominant follicle reaches 17mm or more women will receive Human chorionic gonadotrophin (Choriomon® IBSA, Switzerland) 5000IU and a timed intercourse will be advised 36 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Clomiphene resistant PCOS women

Exclusion Criteria:

* Other causes of infertility.
* Hyperprolactinaemia.
* BMI>35.
* Previous Letrozole or LOD therapy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Ovulation | 6 weeks after starting the intervention
  Regular vaginal ultrasounds will be done at regular intervals starting from the 10th day after the intervention

SECONDARY OUTCOMES:
Pregnancy | 6 months after starting the intervention
  Pregnancy will be diagnosed by the presence of an intra uterine gestational sac during vaginal ultrasound examination one week after a missed period.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] Vendola K, Zhou J, Wang J, Famuyiwa OA, Bievre M, Bondy CA. Androgens promote oocyte insulin-like growth factor I expression and initiation of follicle development in the primate ovary. Biol Reprod. 1999 Aug;61(2):353-7. doi: 10.1095/biolreprod61.2.353. PMID 10411511
- [Background] van Wely M, Bayram N, van der Veen F, Bossuyt PM. Predictors for treatment failure after laparoscopic electrocautery of the ovaries in women with clomiphene citrate resistant polycystic ovary syndrome. Hum Reprod. 2005 Apr;20(4):900-5. doi: 10.1093/humrep/deh712. Epub 2005 Jan 7. PMID 15640254